CLINICAL TRIAL: NCT05275374
Title: A Dose-escalation and Expansion Phase I/IIa Study of XP-102 and XP-102 in Combination With Trametinib in Advanced Solid Tumor Patients With a BRAF V600 Mutation (ENHANCE)
Brief Title: XP-102 and XP-102 in Combination With Trametinib in Advanced Solid Tumor Patients With a BRAF V600 Mutation
Acronym: ENHANCE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XYN-701
Record Dates: First submitted 2022-02-20; First posted 2022-03-11 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cancer; BRAF V600 Mutation; Melanoma; Colorectal Cancer; Thyroid Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Neoplasms; Melanoma; Colorectal Neoplasms; Thyroid Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 - XP-102 Dose Escalation (Experimental): XP-102
  Interventions: Drug: XP-102
- Part 2 - XP-102 + Trametinib Dose Escalation (Experimental): XP-102 plus Trametinib
  Interventions: Drug: XP-102; Drug: Trametinib
- Part 3 - XP-102 + Trametinib Dose Expansion (Experimental): XP-102 plus Trametinib
  Interventions: Drug: XP-102; Drug: Trametinib

INTERVENTIONS:
Drug: XP-102 — XP-102 will be administered orally once or twice daily in a continuous regimen.
Drug: Trametinib — Trametinib will be administered 2mg orally once a day.
  Arms: Part 2 - XP-102 + Trametinib Dose Escalation; Part 3 - XP-102 + Trametinib Dose Expansion

SUMMARY:
This is a first-in-human multi-center study which will be conducted in advanced malignant solid tumors patients. The solid tumor type is limited to melanoma, colorectal, non-small-cell lung, and thyroid cancer with positive BRAF V600 mutation. This study is divided into three stages: Phase Ia: a dose-escalation phase of XP-102; Phase Ib: a dose-escalation and sample size expansion phase of XP-102 plus trametinib; Phase IIa: an expansion phase of XP-102 plus trametinib.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Advanced malignant solid tumor patients with a BRAF V600 mutation (limited to melanoma, colorectal cancer, non-small cell lung cancer, or thyroid cancer).
* Must have failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Prior treatment with BRAF inhibitors and/or MEK inhibitors is permitted；
* At least one measurable lesion (brain metastasis must not be the only measurable lesion) according to Response Evaluation Criteria in Solid Tumours (RECIST v1.1);
* ECOG performance status of 0 or 1;
* Expected survival ≥ 3 months;
* Adequate liver, renal, coagulation, cardiac, and hematologic function.
* A negative pregnancy test if female patient is of reproductive potential.
* For men and women of reproductive potential, agreement to use an effective contraceptive method from the time of screening and throughout their time on study.
* Patients must agree to, and be capable of, adhering to the study visit schedule and all other protocol requirements;
* Patients must understand and voluntarily sign the written informed consent form, before the initiation of any study-specific procedures in the trial.

Exclusion Criteria:

* Active central nervous system (CNS) lesions. However, patients with asymptomatic and brain metastases who received treatment (including targeted brain radiotherapy, surgical treatment, glucocorticoid or other treatments) without disease progression for ≥ 3 months are eligible.
* Patients who received radiotherapy, immunotherapy, hormone therapy, targeted therapy, biotherapy, traditional Chinese medicine therapy, chemotherapy or any clinical trial treatment within 14 days before the first dose.
* Patients who have persistent toxicity caused by previous chemotherapeutic drugs or radiotherapy has not recovered to lower than grade 2 (except hair loss) according to CTCAE version 5.0;
* Patients who are allergic to active substances or excipients of XP-102 or trametinib.
* Significant traumatic injury within 28 days before the first dose of the investigational drug, or if major surgery is anticipated during the course of study treatment;
* According to the judgment of the investigator, patients with dysphagia, or any gastrointestinal diseases that may affect drug absorption or activity;
* Administration of strong inhibitors or inducers of CYP3A4 liver metabolic enzymes within 14 days before the first dose of the investigational drug;
* Patients who are receiving drugs that may prolong QT interval and unable or unwilling to stop treatment or switch to other alternative treatment before study enrollment;
* Symptomatic active fungal, bacterial and/or viral infections; including known HIV, active hepatitis B, active hepatitis C or active syphilis infection.
* Any poorly controlled disorders (such as serious mental, neurological, cardiovascular, respiratory, digestive, urinary, bleeding and coagulation, or other system diseases) that may significantly affect the clinical trial;
* Other situations not suitable for participation in the study as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety of XP-102. | 28 days
  Number of participants with treatment related adverse events.
Evaluate the pharmacokinetics of XP-102. | 28 days
  Blood plasma concentration.
Establish maximum tolerated dose of XP-102. | 28 days
  Number of participants with dose limiting toxicity

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of XP-102 + trametinib. | 28 days
  Blood plasma concentration.
Characterize tolerability of XP-102 in combination with trametinib. | 28 days
  Number of participants with dose limiting toxicity
Evaluate the pharmacokinetics of XP-102 administered with food | 4 days
  Blood plasma concentration.
Evaluate clinical activity/efficacy of XP-102. | Approximately every 8 weeks (up to 2 years)
  Overall Response Rate with RECIST criteria v1.1.

IPD SHARING:
Plan to Share IPD: Undecided